CLINICAL TRIAL: NCT03810885
Title: SalT Reduction InterVEntion: Examination of the Metabolic, Behavioral and Health Consequences of Reducing Salt Intake. A Randomized Controlled Trial in a Real Life Setting
Brief Title: SalT Reduction InterVEntion: Metabolic, Behavioral and Health Consequences of Reducing Salt in Bread
Acronym: STRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Ulla Toft, Associate Professor, PhD, MSc, Head of Section of Health Promotion and Prevention, Bispebjerg Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: H-17030995
Record Dates: First submitted 2018-11-30; First posted 2019-01-22 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Salt Intake
Keywords: 24hr urine collection
MeSH Terms: interventions — Bread; Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Active Comparator:
  Intervention A : Salt reduced bread
  Assigned Interventions: Participants will receive salt reduced bread and no dietary counselling.
  Active Comparator:
  Intervention A+B: Salt reduced bread + Dietary counselling
  Assigned Interventions: Participants in this group will receive both salt reduced bread and dietary counselling to reduce salt and increase potassium intake.
  Placebo comparator:
  Control: normal bread
  Assigned Interventions: Participants will receive bread with a regular content of salt and no dietary counselling.
Who Masked: Participant
Masking Description: The participants will be unaware of the treatment groups and the salt content of the bread products will be blinded to the participants.
  Nurses examining participants at baseline and follow-up will be unaware of which intervention group the families were randomized into. The primary outcome measures will be blinded to the outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Salt reduced bread (Experimental): Bread with reduced salt content
  Interventions: Other: Bread with reduced salt content
- Dietary advice and Salt reduced bread (Experimental): bread with reduced salt content, dietary advice
  Interventions: Other: Bread with reduced salt content; Behavioral: Dietary advice
- Normal bread (Placebo Comparator): Bread with standard salt content
  Interventions: Other: Bread with standard salt content

INTERVENTIONS:
Other: Bread with reduced salt content — Bread with gradually lowered salt content
  Arms: Dietary advice and Salt reduced bread; Salt reduced bread
Behavioral: Dietary advice — Participants will receive information on how to lower salt and increase potassium intake
  Arms: Dietary advice and Salt reduced bread
Other: Bread with standard salt content — Bread with normal salt content
  Arms: Normal bread

SUMMARY:
The trial is conducted as a randomized controlled trial including children and adults recruited as families. The families are randomly allocated into three groups to investigate the effect of different salt reduction strategies in a period of 3-4 months. Families in the first intervention group are receiving salt reduced bread. Families in the second intervention group are receiving salt reduced bread in combination with dietary counselling to reduce salt and increase potassium intake. Families in the control group are receiving bread with a regular content of salt and no dietary counselling.

DETAILED DESCRIPTION:
The trial is conducted as a randomized controlled trial including children and adults recruited as families. The families are randomly allocated into three groups to investigate the effect of different salt reduction strategies in a period of 3-4 months. Families in the first intervention group are receiving salt reduced bread. Families in the second intervention group are receiving salt reduced bread in combination with dietary counselling to reduce salt and increase potassium intake. Families in the control group are receiving bread with a regular content of salt and no dietary counselling.

Participants will be instructed to replace their usual consumption of bread by the bread products provided in the study. In all other respects, participants will be requested to live their lives as usual without changing any habits, except the families receiving dietary counselling. The participants will be unaware of the treatment groups and the salt content of the bread products will be blinded to the participants.

Families will attend a physical examination at baseline and at 3-4 months follow-up. The health examination includes anthropometrics, blood pressure measurements and blood samplings for analysis of glucose, lipid metabolism and hormone balance. Urine samples will be collected to investigate the sodium and potassium content. Furthermore salt-sensitivity and preference tests will be made. After both health examinations the families will collect three repeated 24-hour urine collections at home and fill in a 7 days dietary record.

After data collection, blood and urine samples will be analysed. Analyses from both baseline and follow-up are expected ultimo February 2019, whereby data cleaning and statistical analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Participants living with children
* Adults 18-69 years
* Children 3-17 years
* Daily intake of bread

Exclusion Criteria:

* Diabetes
* Cardiovascular disease
* Antihypertensive treatment
* Lipid-lowering treatment
* Pregnancy
* U-albumin > 300 mg/day
* Celiac disease

Ages: 3 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline sodium level in 24 hour urine at 4 months | Measurements at Baseline and at 4 month.
  Adults average of 3 repeated 24 hour urine, children a single 24hour urine collection; excluding urine first morning including urine of the following morning. Completeness evaluated in adults by Para-Amino-Benzoic-Acid (PABA).

SECONDARY OUTCOMES:
Change from Baseline potassium level in 24 hour urine at 4 months | Measurements at Baseline and at 4 month.
  Adults average of 3 repeated 24 hour urine, children a single 24hour urine collection; excluding urine first morning including urine of the following morning.
Change from Baseline Systolic blood pressure at 4 months | Measurements at Baseline and at 4 month.
  Systolic blood pressure measured at baseline and follow-up . Average of three measurements, with the participant sitting upright at rest.. Minimum 2 hours fasting.
Change from Baseline Diastolic blood pressure at 4 months | Measurements at Baseline and at 4 month.
  Diastolic blood pressure measured at baseline and follow-up . Average of three measurements, with the participant sitting upright at rest.. Minimum 2 hours fasting.
Change from Baseline Adrenaline and Noradrenaline levels in plasma at 4 months | Measurements at Baseline and at 4 month.
  blood sampled, stored on ice, with the participant lying down after 30 minutes of rest. Minimum 2 hours of fasting.
Change from Baseline Renin and Aldosterone levels in plasma at 4 months | Measurements at Baseline and at 4 month.
  blood sampled, with the participant lying down after 30 minutes of rest. Minimum 2 hours of fasting.
Change from Baseline Salt sensitivity and preference at 4 months | Measurements at Baseline and at 4 month.
  Sensory test: Sensitivity and preference test, minimum 2 hours of fasting

OTHER OUTCOMES:
Change from Baseline Glucose levels in plasma at 4 months | Measurements at Baseline and at 4 month.
  blood sampled, with the participant lying down after 30 minutes of rest. Minimum 2 hours of fasting.
Change from Baseline HbA1C levels in full blood at 4 months | Measurements at Baseline and at 4 month.
  blood sampled, with the participant lying down after 30 minutes of rest. Minimum 2 hours of fasting.
Change from Baseline Cholesterol levels in plasma (LDL, HDL, total cholesterol and triglycerides) at 4 months | Measurements at Baseline and at 4 month.
  blood sampled, with the participant lying down after 30 minutes of rest. Minimum 2 hours of fasting.
Change from Baseline Height in centimetres at 4 months | Measurements at Baseline and at 4 month.
  Measured in centimetres to the closest decimal, without shoes or socks, with clothes on
Change from Baseline Weight in kilograms at 4 months | Measurements at Baseline and at 4 month.
  Measured in kilograms to the closest decimal, without shoes or socks, with clothes on
Change from Baseline Impedance in ohm at 4 months | Measurements at Baseline and at 4 month.
  Measured in ohm to the closest decimal, without shoes or socks, with clothes on
Change from Baseline Hip circumference in centimetres at 4 months | Measurements at Baseline and at 4 month.
  Measured on bare skin to nearest decimal
Change from Baseline Waist circumference in centimetres at 4 months | Measurements at Baseline and at 4 month.
  Measured on bare skin to nearest decimal
Baseline Albumin in spot urine | Measurements at Baseline
  Not morning urine, minimum 2 hours of fasting
Change from Baseline Sodium, potassium and creatinine level in spot urine at 4 months | Measurements at Baseline and at 4 month.
  Not morning urine, minimum 2 hours of fasting

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Toft, MSc, PhD, Principal Investigator — Capital Region, Copenhagen, Denmark
Locations (1):
- Center fot Clinical Research and Prevention, Glostrup Municipality, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2017-12-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT03810885/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT03810885/SAP_001.pdf